CLINICAL TRIAL: NCT02964871
Title: Rapid Assessment of and Prophylaxis for Influenza in Dwellers of Long-term Care Facilities
Acronym: Rapid-LTCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1160; A532000 (Other: UW Madison); SMPH\FAMILY MEDICINE (Other: UW Madison)
Record Dates: First submitted 2016-11-07; First posted 2016-11-16 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Influenza, Human; Pneumonia
Keywords: Long-term care facility; Elderly
MeSH Terms: conditions — Influenza, Human; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTCF with RIDT (Active Comparator): Nasal swabs will be tested by nursing personnel at each intervention site using SOFIA Fluorescent Immunoassay Analyzer Influenza A+B (LTCF with RIDT). Anonymous results will be sent, via wireless transmission, for daily review by the study team and public health personnel. A positive influenza detection will trigger direct communication with LTCF personnel with advice on antiviral treatment, antiviral prophylaxis, and appropriate infection control practices. We will collect data from each site regarding the prescribing of influenza antivirals for treatment and prophylaxis, number of hospitalizations, number of deaths, and associated healthcare costs during annual, dynamic, 4-month risk windows, based on Wisconsin surveillance of influenza patterns.
  Interventions: Device: Sofia Fluorescent Immunoassay Analyzer Influenza A+B
- LTCF Control (Placebo Comparator): Usual care.
  Data will be collected from each site regarding the prescribing of influenza antivirals for treatment and prophylaxis, number of hospitalizations, number of deaths, and associated healthcare costs during annual, dynamic, 4-month risk windows, based on Wisconsin surveillance of influenza patterns.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Sofia Fluorescent Immunoassay Analyzer Influenza A+B — The Sofia Influenza A+B Fluorescent Immunoassay (FIA) uses advanced immunofluorescence-based lateral-flow technology to detect influenza A and influenza B viral nucleoprotein antigens.
  Arms: LTCF with RIDT
Other: Usual care — Our team will discuss our interest in monitoring influenza antiviral treatment and prophylaxis courses, antibiotic courses, clinician and emergency room visits, respiratory infection-related hospitalizations, all-cause hospitalizations, and deaths during the anticipated 4-month influenza season over 3 years.
  Arms: LTCF Control

SUMMARY:
RAPID-LTCF is a stratified, block-randomized controlled trial to assess the effectiveness of a simple ARI case definition, rapid influenza diagnostic test (RIDT) with wireless transmission of results, and provision of infection control guidance when influenza is detected. Because of the nature of the intervention, blinding is not possible. Sites will be initially recruited for a study of "respiratory infections within LTCFs." After acceptance into the study, sites will be matched in terms of bed capacity, location, and other features prior to randomization.

DETAILED DESCRIPTION:
Project Overview: The primary goal of RAPID-LTCF is to conduct a randomized, controlled clinical trial (RCT) to assess the effect of on-site, rapid influenza detection at long-term care facilities (LTCFs) on influenza-related hospitalizations, deaths, and healthcare-associated costs.

The basic research question in PICO format is:

Population: for residents of LTCFs across Wisconsin

Intervention: does early detection of influenza coupled with infection control guidance

Comparator: compared to usual care

Outcomes: result in:

1. increase early detection and reporting of influenza outbreaks?
2. increased early antiviral treatment of influenza?
3. increased use of antiviral prophylaxis for other at-risk residents?
4. fewer hospitalizations during the influenza season?
5. reduced mortality during the influenza season?
6. lower healthcare associated costs during the influenza season?

Building on two highly successful pilot QI projects-undertaken during the last two influenza seasons-that confirmed the feasibility and desirability of this approach, existing, CLIA-waived, low-complexity rapid influenza diagnostic test (RIDT) with high sensitivity and high specificity in this population as the diagnostic platform will be used. RIDT analyzers will be configured for wireless transmission of anonymous test results to a cloud-based server for real-time access by public health. Detection of influenza at a LTCF and its transmission to public health in real time will trigger communication and advice on appropriate infection control measures to reduce in-facility transmission. This approach has high potential for limiting influenza's effect at LTCFs.

Residents of LTCFs are at high risk for influenza infection due to reduced efficacy of influenza vaccines in elders, close quartering, presence of co-morbid medical conditions, and delayed response times. Consequently, outbreaks of influenza and other significant respiratory viruses easily spread within LTCFs and cause substantial morbidity and mortality in these populations. Results from this RCT will provide highly generalizable approaches using low-cost, low-complexity and easily-adapted tools and protocols for extremely early influenza detection and response. It is anticipated that early outbreak recognition and control in LTCFs will substantially reduce morbidity, mortality and healthcare associated costs in this vulnerable population.

Background: At present, 1.8 million individuals live in this nation's 16,000 nursing homes and an additional 900,000 live in assisted living facilities. Significant healthcare disparities exist for these individuals; a recent study found that the largest for-profit nursing homes delivered significantly lower quality of care. Part of this disparity is reflected in the fate of those infected with influenza. Influenza and pneumonia combine to form the 8th leading cause of death in the United States. Outbreaks of influenza and other respiratory viruses are common in LTCFs and result in significant morbidity and mortality among residents. This increased morbidity and mortality is due to a combination of close quartering, residents with co-morbid medical conditions, and delays in medical response. Because of this high risk, influenza vaccination has long been recommended for all residents and health care workers in these settings. Influenza vaccines, however, can have very low efficacy in older individuals; vaccine efficacy for protection from the predominant influenza strain in 2014-2015 was estimated to be only 14% for individuals aged 50 years and older. Accordingly, elders (aged 65+) accounted for 72.4% of Wisconsin's influenza-related hospitalizations during the 2014-2015 influenza season and 63% of influenza-related ICU admissions. Moreover, across the country, the rate of attributable influenza hospitalization was 313 per 100,000 for individuals aged 65 year and older.

The current practice for identifying and responding to influenza outbreaks in LTCFs is reactive and delayed. Of 41 known influenza outbreaks in LTCFs during the 2010-2011 season in New York, most were identified retrospectively through reporting of influenza hospitalizations and well before the LTCFs submitted reports to the Department of Health. The availability of CLIA-waived, low-complexity, sensitive and specific rapid influenza detection tests (RIDTs) can facilitate on-site diagnosis and early detection of an outbreak. Coupling RIDTs with wireless transmission of anonymous results directly to public health officials provides the means for extremely early and proactive outbreak recognition and intervention.

Program Goal: A randomized, controlled clinical trial to assess the effect of on-site RIDTs at LTCFs on subsequent influenza-related hospitalizations, deaths, and healthcare-associated costs is proposed. LTCF nursing staff will use RIDT technology to screen residents with acute respiratory infections (ARI). The proposed RIDT is a CLIA-waved, low-complexity test that uses a benign nasal swab specimen. It is configured to send test results via wireless transmission to a cloud platform. From there, data can be accessed in real-time by public health partners.

Methods: Starting in January 2013, extensive experience with the Quidel SOFIA Influenza A+B system at 20 clinical sites and 7 LCTFs where the testing platform transmits influenza test results immediately to a cloud-based system with public health access has been acquired. True "real-time" availability of surveillance results are achievable. Since initiation, this highly innovative system has been working flawlessly. A plan to conduct RAPID-LTCF over three sequential influenza seasons to adapt to the uncertainties of influenza epidemiology has been proposed. Twenty LTCFs across Wisconsin will be recruited for participation and randomized, following stratification, to intervention (RIDT) or control (usual care) arms. Waived consent for on-site specimen collection from residents at the RIDT sites with acute respiratory infections has been approved by the IRB. Nasal swabs will be tested by nursing personnel at each intervention site using SOFIA. Anonymous results will be sent, via wireless transmission, for daily review by the study team and public health personnel. A positive influenza detection will trigger direct communication with LTCF personnel with advice on antiviral treatment, antiviral prophylaxis, and appropriate infection control practices. Data will be collected from each site regarding the number of courses of influenza antiviral medication provided for influenza treatment and for influenza prophylaxis, number of hospitalizations, number of deaths, and associated healthcare costs during annual, dynamic, 4-month risk windows, based on Wisconsin surveillance of influenza patterns. An independent data monitoring and safety board will continuously review outcomes and halt the study should significant differences between the two arms emerge. Outcomes will be assessed using standard statistical methods.

Significance: This program reflects the full intent of the Wisconsin Partnership Program and the Wisconsin Idea by identifying high-risk populations, and combining research, education and public health practice to reduce the disparities of care experienced by these populations. The application of cutting-edge, inexpensive, high-performing and reliable technology into a population of traditionally under-served, high-risk individuals would provide a translatable model for very early and proactive detection of, and response to influenza in LTCFs, thus allowing for appropriate medical (antiviral) and public health (in-room quarantining, enhanced personal protection equipment, prophylaxis of other residents) interventions.

ELIGIBILITY:
Inclusion Criteria:

* Any resident of one of the 10 LTCF intervention facilities with two acute respiratory infection symptoms (rhinorrhea/runny nose, nasal congestion, sore throat, cough or fever).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of influenza antiviral treatment courses provided during the 4-month influenza seasons in RAPID-LTCF vs. control LTCF | 4 months
  Oseltamivir is the most commonly used antiviral for influenza treatment. The usual dose is 75 mg twice a day for 5 days.
Number of influenza antiviral prophylaxis courses provided during the 4-month influenza season in RAPID-LTCF vs. control LTCF | 4 months
  Oseltamivir is the most commonly used antiviral for influenza prophylaxis. The usual dose is 75 mg daily for the duration of likely exposure
Number of respiratory infection-related hospitalizations in RAPID-LTCF vs control LTCF during the 4-month influenza season | 4 months
  These will include all hospitalizations that include a discharge diagnosis for any respiratory infection.
Number of all-cause hospitalizations in RAPID-LTCF vs. control LTCF during the 4-month influenza season | 4 months
  All transfers of patients to the hospital will be assessed.
Deaths during the 4-month influenza season in RAPID-LTCF vs. control LTCF | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon Temte, MD PhD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: Undecided